CLINICAL TRIAL: NCT01008397
Title: Phase 1 Study of AHIST in Seasonal Allergic Rhinitis Patients
Brief Title: Study of AHIST in Seasonal Allergic Rhinitis Patients
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Manufacturer unable to produce
Sponsor: Magna Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHIST IND
Record Dates: First submitted 2009-10-27; First posted 2009-11-05 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2011-02

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Rhinitis, Allergic, Seasonal
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AHIST for seasonal allergic rhinitis (Experimental): AHIST for SAR: each green tablet contains 12mg chlorpheniramine tannate.
  Interventions: Drug: AHIST NDC#58407-012-01

INTERVENTIONS:
Drug: AHIST NDC#58407-012-01 — Oral tablet containing chlorpheniramine tannate 12mg.

SUMMARY:
Objectives:

A) To gather pharmacodynamic measurements and assess blood levels of the active ingredients in AHIST over the dosage interval period of 12 hours.

Hypothesis: Hysteresis curves plotting each active ingredient's blood levels over a 12-hour dosage interval will substantiate S5 Symptom Diary scores (IE: evidentiary therapeutic window data);

B) To report subjective scores by subjects rating the efficacy of a single dose AHIST in relieving nasal congestion, rhinorrhea, nasal itching, sneezing, and post-nasal drip over a 12-hour dosage interval.

Hypothesis: Greater than 66% of subjects will document clinically significant relief over a 12-hour period from one dose of AHIST;

C) Report any side effects or adverse drug reactions and rate the severity of any incidence.

Hypothesis: Not more than one patient will have an adverse event significant enough to warrant withdrawal; side effects will be mild with the most frequently reported side effect occurring in less than 10% of patients-drowsiness.

DETAILED DESCRIPTION:
This Phase 1 clinical trial will be a single dose pharmacokinetics study comprised of 21 individuals with five blood draws over a 12 hour period. Additionally, subjects will subjectively score symptom relief and report any side effects from the single dose of AHIST. Schulman Associates Institutional Review Board (Cincinnati, OH) will approve the study protocol and statement of informed consent. Each study participant will give written informed consent (See Attachment A). Safety will be assured through close observation and physical examination of subjects before, during and at study conclusion. This interventional study will be conducted during the spring allergy season of 2010.

MAGNA plans to show that chlorpheniramine tannate is a safe and effective B.I.D. drug treatment regimen, "indicated for the relief of symptoms associated with seasonal allergic rhinitis in adults and children 12 years of age and older. Treated symptoms include nasal congestion, sneezing, rhinorrhea, itchy nose, itchy/watery eyes, and post nasal drip syndrome [reduction in tickly cough (acute or chronic), mucus in the back of the throat, sore throat, and hoarseness]."

ELIGIBILITY:
Inclusion Criteria:

1. Male and females of any ethnic group between 18 and 60 years of age.
2. History of moderate to severe Seasonal Allergic Rhinitis (SAR) for at least two years.
3. Subjects' symptoms resulting from the irritation of sinus, nasal and upper respiratory tract tissues will include the five symptoms ("S5") that are the focus of this study: nasal congestion, rhinorrhea, nasal itching, sneezing, and post nasal drip.
4. Prior to study drug administration, subjects' good health will be confirmed by medical history, physical examination, and urine dip pregnancy test.
5. Allergic hypersensitivity will be confirmed by an appropriate test as deemed necessary by the physician or well established patient medical history.

Exclusion Criteria:

1. Pregnancy or lactation.
2. Immunotherapy unless at stable maintenance dose.
3. Presence of a medical condition that might interfere with treatment evaluation or require a change in therapy including but not limited to high blood pressure or urinary retention problems.
4. Alcohol dependence.
5. Use of any other investigational drug in the previous month.
6. Subjects presenting with asthma requiring corticosteroid treatment.
7. Subjects with multiple drug allergies.
8. Subjects known to have an idiosyncratic reaction to any of the ingredients in AHIST.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2011-04 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
To gather pharmacodynamic measurements and assess blood levels (five draws) of the active ingredient in AHIST over the dosage interval period of 12 hours. | April 2011

SECONDARY OUTCOMES:
To report any side effects or adverse drug reactions and rate the severity of incidence. | April 2011

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Pollard, MD, Principal Investigator — Family Allergy and Asthma Research Institute
Locations (1):
- Family Allergy and Asthma Research Institute, Louisville, Kentucky, United States